CLINICAL TRIAL: NCT01148901
Title: Hip Arthritis Associated With AS Efficacy and Safety of Early Treatment With Infliximab (Remicade®)
Brief Title: Effectiveness and Safety of Early Treatment With Infliximab for Hip Arthritis Associated With Ankylosing Spondylitis (AS) (P06451)
Acronym: HACER
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No patient enrolled after 6 months from the start. The decision to withdraw the study was based on a feasibility reevaluation conducted with investigators.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Hospital Universitario Reina Sofia de Cordoba (Other Government); Dr. Jose María Martos Becerra (Central Radiological Assessment) - Hospital de Alta Resolución, Puente Genil (Spain) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P06451; 2009-016587-36 (EudraCT Number)
Record Dates: First submitted 2010-06-21; First posted 2010-06-22 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing spondylitis; Hip arthritis; Infliximab
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Remicade (Experimental): Infliximab 5 mg/kg was administered as specified in the Summary of Product Characteristics for patients with ankylosing spondylitis
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — Infliximab 5 mg/kg administered as an intravenous perfusion over a period of 2 hours at Weeks 0, 2, 6, and 14, as indicated in the Summary of Product Characteristics
  Other Names: Remicade, SCH 215596

SUMMARY:
This trial is designed to measure improvement of hip involvement in patients with ankylosing spondylitis (AS) after receiving 4 doses of infliximab. Participants will receive infliximab 5 mg/kg (as an intravenous perfusion over a period of 2 hours) at Weeks 0, 2, 6, and 14, consistent with the approved dosing regimen described in the label. Participants will be evaluated for hip pain, functional capacity and stiffness before and after 14 weeks (4 doses) of treatment. Further treatment after 4 doses is based on standard clinical practice as determined by the trial site.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Ankylosing spondylitis (AS) diagnosis
* Have all 3 of the following:
* Presence of hip pain (nocturnal inflammatory pain)
* Limitation of hip mobility
* Patient's Global Assessment Visual Analog Scale (0-10 cm) ≥4 cm.
* Inadequate response or intolerance to non-steroidal anti-inflammatory drugs (NSAIDs)
* Eligible to be treated with Infliximab (Remicade®)

Exclusion Criteria:

* Causes of coaxalgia other than coxitis of AS, demonstrated by images or laboratory tests
* Women who are pregnant or nursing or plan to nurse or become pregnant
* Serious infections like sepsis, abscesses.
* History of or current certain infections
* History of or current certain medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with clinical improvement assessed by the Western Ontario and McMaster University Osteoarthritis Index (WOMAC) questionnaire | Baseline and Week 15